CLINICAL TRIAL: NCT07404683
Title: Safety, Utility and Effects After 8 Weeks of High-intensity Strength Training With Blood Flow Restriction in the Rotator Cuff
Brief Title: Safety and Effects of High-Intensity Blood Flow Restriction Training in the Rotator Cuff
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Adrián Escriche Escuder, Assistant professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-FIS-4211701
Record Dates: First submitted 2026-02-02; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy Adult
Keywords: blood flow restriction; exercise; high-intensity; rotator cuff
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-intensity exercise with blood occlusion (Experimental): Sixteen sessions of exercise during 8 weeks, 70% repetition maximum, and 50% blood occlusion
  Interventions: Device: High-intensity exercise with BFR
- Low-intensity exercise with blood occlusion (Active Comparator): Sixteen sessions of exercise during 8 weeks, 30% repetition maximum, and 50% blood occlusion
  Interventions: Device: Low-intensity exercise with BFR
- High-intensity exercise without blood occlusion (Active Comparator): Sixteen sessions of exercise during 8 weeks, 70% repetition maximum, without blood occlusion
  Interventions: Procedure: High-intensity exercise without BFR

INTERVENTIONS:
Device: High-intensity exercise with BFR — Three exercises: external rotation at 0°, internal rotation at 0° and elevation in the scapular plane. 4 sets (30, 15, 15, reps to fatigue) with a intensity of 70% RM and a 50% of arterial occlusion pressure. 30" rest between sets, 2' rest between exercises.
  Arms: High-intensity exercise with blood occlusion
Device: Low-intensity exercise with BFR — Three exercises: external rotation at 0°, internal rotation at 0° and elevation in the scapular plane. 4 sets (30, 15, 15, reps to fatigue) with a intensity of 30% RM and a 50% of arterial occlusion pressure. 30" rest between sets, 2' rest between exercises.
  Arms: Low-intensity exercise with blood occlusion
Procedure: High-intensity exercise without BFR — Three exercises: external rotation at 0°, internal rotation at 0° and elevation in the scapular plane. 4 sets (30, 15, 15, reps to fatigue) with a intensity of 70% RM and a without flow restriction application (cuff applied without pressure). 30" rest between sets, 2' rest between exercises.
  Arms: High-intensity exercise without blood occlusion

SUMMARY:
This study aims to analyze the effects of an 8-week strength training program combining different exercise intensities and blood flow restriction (BFR) conditions on safety, tolerability, muscle adaptations, and physical performance variables. Three training modalities will be compared: 1) high-intensity exercise with BFR therapy; 2) low-intensity exercise with BFR therapy; and 3) high-intensity exercise without BFR therapy. All groups will perform the same exercise modality, differing only in intensity and the application of BFR.

Participants will be randomly assigned to one of the three groups and will undergo a 8-week intervention. The variables of interest will be assessed in each group for subsequent analysis and comparison.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, untrained adults
* Age between 18 and 65

Exclusion Criteria:

* Current participation in an upper limb strength training program
* Presence of comorbidities that increase cardiovascular risk (uncontrolled ischemic heart disease, uncontrolled hypertension, diabetes, etc.)
* Patients with more than one thromboembolism risk factor (obesity, history of thrombosis, prolonged immobilization, recent surgery, use of contraceptives, etc.)
* Current diagnosis of any pathology affecting the cervical spine, shoulder, and/or thoracic spine
* History of surgery in the last year
* Use of ergogenic aids or medications that affect muscle metabolism (anabolic steroids, testosterone, creatine, protein supplements, corticosteroids, chronic use of nonsteroidal anti-inflammatory drugs, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Isometric rotator cuff strength | Baseline, 4 weeks and 8 weeks
  Isometric rotator cuff strength measured with a dynamometer
Rate of perceived exertion | Periprocedural
  Rate of perceived exertion (RPE) measured using the Borg scale (0-10)
Perceived tolerance | 8 weeks
  Participant tolerance to the training protocol will be assessed at the end of the intervention using a 5-point Likert scale, ranging from very well tolerated (5), well tolerated (4), neutral (3), poorly tolerated (2), to very poorly tolerated (1).
Occurrence of adverse effects | Immediately after the intervention, 1 hour, 6 hours, 24 hours, 1 week
  Occurrence of adverse effects (e.g., pain, delayed onset muscle soreness, sudden weakness of the trained limb, redness or swelling of the trained limb, etc.) by self-report
Surface electromyography | Periprocedural
  Surface electromyography for the study of muscle recruitment (middle deltoid, infraspinatus, teres minor and trapezius muscles)
Muscle Thickness | Baseline, 4 weeks, 8 weeks
  Muscle thickness of the deltoid, biceps brachii, triceps brachii, and pectoralis major will be assessed using ultrasound imaging

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Escriche-Escuder, PhD, Principal Investigator — University of Valencia

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study will be available from the corresponding author upon reasonable request.